CLINICAL TRIAL: NCT02718079
Title: High-Volume Plasma Exchange Versus Standard Medical Treatment in Patients With Acute Liver Failure-A Prospective Randomized Pilot Trial
Brief Title: High-Volume Plasma Exchange Versus Standard Medical Treatment in Patients With Acute Liver Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ALF-03
Record Dates: First submitted 2016-02-29; First posted 2016-03-24 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Acute Liver Failure
MeSH Terms: conditions — Liver Failure, Acute | interventions — Plasma Exchange; Intubation, Intratracheal; Sodium Chloride; Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard medical therapy with Plasma Exchange (Experimental): Plasma Exchange will be performed for consecutive days. Standard medical therapy included as per requirement,management of cerebral edema/intracranial hypertension: transfer to ICU,prophylactic antibiotics, intubation of trachea (as required),administration of mannitol or 3% saline for severe elevation of Intra Cranial Pressure,volume replacement and pressor support (norepinephrine, vasopressin) as needed, NAC, correction of metabolic parameters and nutrition.
  Interventions: Biological: Plasma Exchange; Other: Management of cerebral edema/intracranial hypertension:; Other: Transfer to Intensive Care Unit; Drug: Prophylactic Antibiotics; Other: Intubation of trachea; Other: Administration of mannitol or 3% saline for severe elevation of Intra Cranial Pressure; Other: Volume Replacement; Other: Pressor Support; Drug: N-acetyl-L-cysteine; Other: Correction of metabolic parameters; Dietary Supplement: Correction of nutrition
- Standard medical therapy alone (Active Comparator): Standard medical therapy included as per requirement,management of cerebral edema/intracranial hypertension: transfer to ICU,prophylactic antibiotics, intubation of trachea (as required),administration of mannitol or 3% saline for severe elevation of Intra Cranial Pressure,volume replacement and pressor support (norepinephrine, vasopressin) as needed, NAC, correction of metabolic parameters and nutrition.
  Interventions: Other: Management of cerebral edema/intracranial hypertension:; Other: Transfer to Intensive Care Unit; Drug: Prophylactic Antibiotics; Other: Intubation of trachea; Other: Administration of mannitol or 3% saline for severe elevation of Intra Cranial Pressure; Other: Volume Replacement; Other: Pressor Support; Drug: N-acetyl-L-cysteine; Other: Correction of metabolic parameters; Dietary Supplement: Correction of nutrition

INTERVENTIONS:
Biological: Plasma Exchange
  Arms: Standard medical therapy with Plasma Exchange
Other: Management of cerebral edema/intracranial hypertension:
Other: Transfer to Intensive Care Unit
Drug: Prophylactic Antibiotics
Other: Intubation of trachea
Other: Administration of mannitol or 3% saline for severe elevation of Intra Cranial Pressure
Other: Volume Replacement
Other: Pressor Support
Drug: N-acetyl-L-cysteine
Other: Correction of metabolic parameters
Dietary Supplement: Correction of nutrition

SUMMARY:
The study will be conducted on patients admitted to Department of Hepatology from Jan 2016 to Jan 2018 at Institute of Liver & Biliary Sciences, New Delhi. Study group will comprise of patients with acute liver failure (ALF) who have no option for liver transplant (due to any reason) or have contraindications for liver transplant or have no prospective living donor and will be assessed for enrollment in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute liver failure defined as : Patients with jaundice which is complicated by encephalopathy and coagulopathy within 4 weeks of the onset of jaundice and without underlying chronic liver disease.

Exclusion Criteria:

* Age <12 or > 75 years
* Hepato-Cellular Carcinoma
* Active untreated Sepsis/DIC
* Any evidence of active bleed secondary to coagulopathy
* Hemodynamic instability requiring high dose of Vasopressors
* Coma of non-hepatic origin.
* Pregnancy
* Comorbidities associated with poor outcome (Extrahepatic neoplasia, severe cardiopulmonary disease defined by a New York Heart Association score >3, or oxygen/steroid-dependent chronic obstructive pulmonary disease).
* Patients being taken up for liver transplant
* Refusal to participate in the study.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Survival in both groups. | 21 days

SECONDARY OUTCOMES:
Duration of Intensive Care Unit stay in both groups. | 21 days
Improvement in SIRS (Systemic Inflammatory Response Syndrome) score. | 48 hours
Improvement in SIRS (Systemic Inflammatory Response Syndrome) score. | day 5
Improvement in SIRS (Systemic Inflammatory Response Syndrome) score. | day 7
Improvement in SOFA (Sequential Organ Failure Assessment) score. | 48 hours
Improvement in SOFA (Sequential Organ Failure Assessment) score. | day 5
Improvement in SOFA (Sequential Organ Failure Assessment) score. | day 7
Improvement in APACHE II (Acute Physiology and Chronic Health Evaluation) score. | 48 hours
Improvement in APACHE II (Acute Physiology and Chronic Health Evaluation) score. | Day 5
Improvement in APACHE II (Acute Physiology and Chronic Health Evaluation) score. | Day 7
Effect on systemic haemodynamics in both groups. | 24 hours
  Effect is defined as resolution of SIRS (Systemic Inflammatory Response Syndrome).
Effect on systemic haemodynamics in both groups. | 48 hours
  Effect is defined as resolution of SIRS (Systemic Inflammatory Response Syndrome).
Pro inflammatory cytokines profile in both groups. | 1 hour
Serum Endotoxin levels in both groups. | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Dr Rakhi Maiwall, DM, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maiwall R, Bajpai M, Singh A, Agarwal T, Kumar G, Bharadwaj A, Nautiyal N, Tevethia H, Jagdish RK, Vijayaraghavan R, Choudhury A, Mathur RP, Hidam A, Pati NT, Sharma MK, Kumar A, Sarin SK. Standard-Volume Plasma Exchange Improves Outcomes in Patients With Acute Liver Failure: A Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2022 Apr;20(4):e831-e854. doi: 10.1016/j.cgh.2021.01.036. Epub 2021 Jan 29. PMID 33524593